CLINICAL TRIAL: NCT05797935
Title: Evaluation of Changes in Pancreatic Fat Content Using Advanced MR Sequences in Diabetics on Dapagliflozin Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ashu Rastogi, Associate professor, Department of endocrinology and metabolism , PGIMER chandigarh, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 9805821254
Record Dates: First submitted 2023-03-22; First posted 2023-04-04 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Pancreatic Lipomatosis
Keywords: Dapagliflozin; Pancreatic fat; MRI; Diabetes; MRS
MeSH Terms: conditions — Diabetes Mellitus | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Randomised Control Trial
Who Masked: Investigator
Masking Description: Single blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (No Intervention): Only the standard drugs for type 2 diabetes were given. Dapagliflozin was not given in this group.
- Dapagliflozin group (Active Comparator): The patients were given standard drugs for type 2 diabetes and Dapagliflozin.
  Interventions: Drug: Dapagliflozin 10mg Tab

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — Dapagliflozin was given at a dose of 10 mg/day in one group and its effect was observed on the pancreatic fat content
  Arms: Dapagliflozin group

SUMMARY:
The study aimed to assess changes in pancreatic fat content in people with diabetes on dapagliflozin (SGLT2 inhibitor) and beta cell function.

DETAILED DESCRIPTION:
The study assessed and estimated the difference in pancreatic fat content in the patients of Type 2 Diabetes Mellitus at baseline and after taking dapagliflozin for 24 weeks.

The investigators even estimated the correlation between two advanced MR techniques commonly used for quantification of pancreatic fat (PDFF and MR Spectroscopy)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years,
2. Hba1c 7-11%,
3. Renal function (MDRD) > 30 ml/min, on glucose-lowering therapy {metformin, sulfonylureas, glinides, dipeptidyl peptidase-4 (DPP-4) inhibitors, or basal insulin} at a stable dose for at least 3 months.

Exclusion Criteria:

1. Uncontrolled hyperglycemia at screening (fasting blood glucose FBG ≥ 240 mg/dL).
2. Diabetes other than type 2 diabetes
3. Age younger than 18 years.
4. Pregnant patients or lactating.
5. Patients who refuse to give consent to be enrolled in the study.
6. Any contraindication to magnetic resonance imaging.
7. More than 5% total body weight loss within the last month.
8. Patients with moderate or severe renal impairment
9. Any contraindication to SGLT2i
10. Prior SGLT2i within the past 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
To assess and estimate the difference in pancreatic fat content in the patients of Type 2 Diabetes Mellitus at baseline and after taking dapagliflozin for 24 weeks | 24 weeks
  The pancreatic fat percentage will be measured by MRI sequences at baseline and at 24 weeks and a change will be compared

SECONDARY OUTCOMES:
To estimate the correlation between two advanced MR techniques commonly used for quantification of pancreatic fat(PDFF and MR Spectroscopy) | 24 weeks
  The pancreatic fat percentage will be measured by MRI sequences at baseline and at 24 weeks and a correlation will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Deptt of Endocrinology, Chandigarh, India